CLINICAL TRIAL: NCT00668824
Title: Improved Diagnosis of Congenital Heart Disease by Magnetic Resonance Imaging Using Vasovist
Acronym: CHD Vasovist
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guy's Hospital (Other)
Responsible Party: Jackie Pullen, King's College London
Purpose: Diagnostic
Other Study IDs: 07/Q0704/2; ISRCTN23698917
Record Dates: First submitted 2008-04-24; First posted 2008-04-29 (Estimated); Last update posted 2009-08-03 (Estimated); Status verified 2009-07

CONDITIONS: Congenital Heart Disease
Keywords: Congenital Heart Disease (CHD)
MeSH Terms: conditions — Heart Defects, Congenital | interventions — gadofosveset trisodium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Vasovist

SUMMARY:
Magnetic Resonance Imaging (MRI) is an effective and radiation free method of diagnosing Congenital Heart Disease (CHD). MRI works by taking images of the anatomy and physiology. These images also provide information on the hearts function and blood flow. The clarity of these images is enhanced by the use of contrast agents (dyes). However these agents only stay in the blood vessels for a short time and therefore limit the time in which the better quality images can be obtained. This study aims to determine whether MRI using Vasovist (a dye that stays in the vessels for a prolonged period of time) can improve the diagnosis of Congenital Heart Disease (CHD) by allowing more areas to be imaged and the improved assessment of various parameters (anatomy, volumes, flow) as well as vastly improving image quality.

DETAILED DESCRIPTION:
We planned an intra-individual study, where 20 adult patients with CHD (e.g. Fallot Tetralogy, s/p corrective surgery, single ventricle s/p Fontan operation, aortic and pulmonary artery stenosis) will undergo two examinations. Both scans are aimed to assess different diagnostic parameter like angiography, cardiac anatomy, ventricular volume and flow.

The first clinically indicated scan in our clinically established imaging protocol is performed using a standard contrast agent. The second scan is performed using a new protocol with Vasovist within the next seven days. Informed consent for the additional second scan will be obtained. In order to optimise the scan protocol for Vasovist we plan a pilot phase using three patients. Dosage of the two contrast agents will be within the approved dose. Any adverse events will be immediately reported. The following diagnostic parameters will be assessed and compared between standard Gadolinium (Gd) agent and Vasovist.

1. MR-Angiography (MRA): assessment of the MRA quality of the large systemic and the pulmonary vessel (arterial and venous) by measuring the Contrast-to-Noise Ratio (CNR) and the vessel sharpness. In addition, the overall image-quality will be scored by three independent readers (scale: excellent, good, ok, bad).
2. Cardiac Anatomy: assessment of image quality of the cardiac anatomy from 3D single/dual phase MRI by measuring Signal-to-Noise Ratio (SNR) and CNR as well as assessing the overall image quality by three independent readers (scale: excellent, good, ok, bad).
3. Ventricular Volumes: comparison of systolic and diastolic volumes measured from multi-slice 2D short axis cine MRI, two single phases 3D whole heart MRI (diastole and systole).
4. Flow: the different flow values will be measured in the large vessels using the Phase Contrast Angio (PCA) data. Furthermore, the flow reproducibility will be determined by using two scans. The overall scan-time to assess all these parameter will be approximately 40 minutes. The intra-individual study allows a direct comparison of the different parameters in a number of vascular territories.

ELIGIBILITY:
Inclusion Criteria:

* The main inclusion criteria will be patient with CHD, i.e. complex congenital defects such as:

  1. Aortic abnormalities
  2. Pulmonary artery abnormalities
  3. Systemic or pulmonary venous abnormalities
  4. The study will be limited to patients aged 18 and over

Exclusion Criteria:

* The study will involve MR contrast agents and and MRI scans, therefore the principle exclusion criteria are:

  1. Any contra-indications to MR (e.g. pacemakers)
  2. Known allergy to MR contrast agents
  3. Patients not agreeing to take part in study
  4. Pregnancy and nursing mothers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2007-03; Primary Completion 2008-07 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
The improvement of diagnosis of CHD, due to larger coverage of vascular territories, higher spatial resolution, faster acquisition and higher quality of MR-flow measurements using Vasovist in comparison with standard Gd-agent
The improvement of image quality will be analysed by measuring the SNR, the CNR, the vessel sharpness. In addition, the overall image quality will be scored by three independent readers (scale: excellent, good, ok, bad)
Ventricular volumes measured from the acquired data will be compared with respect to a reference
The accuracy (standard deviation) and reproducibility of the flow measurements will be compared using the two different agents

SECONDARY OUTCOMES:
No secondary outcome measures.

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Imaging Sciences, London, United Kingdom